CLINICAL TRIAL: NCT05800964
Title: Phase 1 First-In-Human Study to Explore the Safety, Tolerability, and Pharmacokinetics of AMG 305 in Subjects With Advanced Solid Tumors
Brief Title: Study to Explore the Safety, Tolerability, and Pharmacokinetics of AMG 305 in Subjects With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20220073; 2022-502867-39 (EudraCT Number)
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
Keywords: Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Dose Exploration (Experimental): Participants will receive escalating doses of AMG 305.
  Interventions: Drug: AMG 305
- Part B: Dose Expansion (Experimental): Participants with selected solid tumors will receive the RP2D identified in Part A.
  Interventions: Drug: AMG 305

INTERVENTIONS:
Drug: AMG 305 — Short-term intravenous (IV) infusion

SUMMARY:
The primary objective of this study is to:

* Evaluate the safety and tolerability of AMG 305 in adult participants
* Determine the optimal biologically active dose (OBD), at or below the maximum tolerated dose (MTD) with MTD 1 as the maximum tolerated starting dose and MTD 2 as the maximum tolerated target dose
* Determine the recommended phase 2 dose (RP2D)

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has provided informed consent to the main study prior to initiation of any study specific activities/procedures
* Male or female participants age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Participants with histologically or cytologically documented selected solid tumor diseases. Participants must have exhausted available standard of care (SOC) systemic therapy or must not be candidates for such available therapy
* For dose expansion cohorts: participants with at least 1 measurable lesion ≥10 mm which has not undergone biopsy within 3 months of screening scan. This lesion cannot be biopsied at any time during the study
* Life expectancy > 3 months
* Adequate organ function

Key Exclusion Criteria:

* Untreated central nervous system (CNS) metastases, leptomeningeal disease, or spinal cord compression
* History of other malignancy within the past 2 years
* Ongoing or active infection (including chronic or localized)
* Any pleural effusion or pericardial effusion within 4 weeks or ascites requiring recurrent drainage procedures or other medical intervention within 2 weeks prior to the first dose of the investigational products.
* Known interstitial lung disease
* Positive test for human immunodeficiency virus (HIV)
* Positive hepatitis B surface antigen or positive hepatitis C virus ribonucleic acid (RNA) by polymerase chain reaction (PCR)
* History of non-infectious/immune-checkpoint inhibitor related pneumonitis that required corticosteroids, or current or suspected pneumonitis that cannot be ruled out by imaging at screening.
* Anticancer therapies including radiotherapy (with the exception of palliative radiation) chemotherapy or molecularly targeted treatments or tyrosine kinase inhibitors (TKI) within 4 weeks of administration of the first dose of AMG 305; checkpoint inhibitor therapy within 3 months of the first dose of AMG 305; or other immunotherapies/monoclonal antibodies within 3 weeks of administration of the first dose of AMG 305.
* Has had a major surgery within 4 weeks of administration of a first dose of study treatment
* Autoimmune disorders requiring chronic systemic steroid therapy or any other form of immunosuppressive therapy while on study (eg, ulcerative colitis, Crohn's disease)
* Live and/or live-attenuated vaccines received within 28 days (or longer, if required locally) prior to the first dose of AMG 305
* Participants with unresolved toxicities from prior anti-tumor therapies to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1 or better, with the exception of alopecia and grade 2 peripheral neuropathy, which has been unchanged within the last 2 months and there is agreement to allow by both the investigator and sponsor
* Currently receiving treatment in another investigational device or drug study
* Female participants of childbearing potential or male participants unwilling to use protocol specified method of contraception
* Females who are pregnant, breastfeeding or who plan to breastfeed or become pregnant while on study
* History or evidence of any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Experience Dose Limiting Toxicities (DLTs) | Day 1 to Day 28
Percentage of Participants who Experience Treatment-Emergent Adverse Events (TEAEs) | Up to a maximum of 2 years
  Adverse events (AEs) are defined as any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are any event that occurs after the participant has received study treatment. Any clinically significant changes in vital signs, electrocardiograms (ECGs), and clinical laboratory tests, as assessed by the investigator, will also be reported as TEAEs.
Percentage of Participants who Experience Treatment-Related Adverse Events | Up to a maximum of 2 years

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of AMG 305 | Up to a maximum of 2 years
Minimum Serum Concentration (Cmin) of AMG 305 | Up to a maximum of 2 years
Area Under the Concentration-Time Curve (AUC) of AMG 305 | Up to a maximum of 2 years
Objective Response Rate (ORR) based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | Up to a maximum of 2 years
  ORR is defined as best overall response (BOR) of complete response (CR) or partial response (PR), Clinical Benefit Rate (defined as BOR of CR, PR, or stable disease [SD] with duration of 24 weeks or longer) based on RECIST v1.1.
ORR based on Immune Response Evaluation Criteria in Solid Tumors (iRECIST) | Up to a maximum of 2 years
  ORR is defined as immune best overall response (iBOR) of immune complete response (iCR) or immune partial response (iPR), Clinical Benefit Rate (defined as iBOR of iCR, iPR, or immune stable disease [iSD] with duration of 24 weeks or longer) based on iRECIST.
Duration of Response (DOR) | Up to a maximum of 2 years
  DOR is defined as the time from the first documentation of objective response until the first documentation of disease progression or death due to any cause, whichever occurs first) by RECIST v1.1 and iRECIST.
Time to Progression | Up to a maximum of 2 years
  Time to progression is defined as the time rom first AMG 305 dose until the first documentation of radiological disease progression by RECIST v1.1 and iRECIST.
Progression-Free Survival (PFS) | Up to a maximum of 2 years
  PFS is defined as the time from first AMG 305 dose until the first documentation of radiologic disease progression or death due to any cause, whichever occurs first) by RECIST v1.1 and iRECIST.
Overall Survival (OS) at 1 Year | 1 year
OS at 2 Years | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (27):
- United States (6):
  - City of Hope National Medical Center, Duarte, California
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York University Cancer Institute, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Next Oncology, San Antonio, Texas
- Australia (2):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- France (2):
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Germany (3):
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Wuerzburg, Würzburg
- National Cancer Center Hospital East, Kashiwa-shi, Chiba, Japan
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
- United Kingdom (6):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Sarah Cannon Research Institute UK, London
  - University College London Hospital, London
  - Christie Hospital, Manchester
  - Freeman Hospital, Newcastle
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com